CLINICAL TRIAL: NCT02279563
Title: A Randomized, Double-blind, Placebo-controlled,Parallel-group Study Comparing the Bioequivalence of Azelastine Hydrochloride and Fluticasone Propionate Nasal Spray (Apotex, Inc.) to That of Dymista™ Nasal Spray (Meda Pharmaceuticals, Inc. )in the Treatment of Seasonal Allergic Rhinitis
Brief Title: A Study Comparing the Bioequivalence of Azelastine Hydrochloride and Fluticasone Propionate Nasal Spray (Apotex, Inc.) to That of Dymista™ Nasal Spray (Meda Pharmaceuticals, Inc.) in the Treatment of Seasonal Allergic Rhinitis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Apotex Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AZFL-NASU-05RB02-CE
Record Dates: First submitted 2014-10-28; First posted 2014-10-31 (Estimated); Last update posted 2014-10-31 (Estimated); Status verified 2014-10

CONDITIONS: Seasonal Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal | interventions — azelastine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Azelastine HCl and Fluticasone Propionate Nasal Spray (Experimental): The investigational product was administered via nasal inhalation with one spray in each nostril twice daily.
  Batch Number KL1981, Expiry Date Mar 2015.
  Interventions: Drug: Azelastine HCl and Fluticasone Propionate Nasal Spray, 137 µg/50 µg per spray
- Dymista™ Nasal Spray (Active Comparator): The reference product was administered via nasal inhalation with one spray in each nostril twice daily.
  Batch Number G30349, Expiry Date Mar 2015.
  Interventions: Drug: Dymista™ Nasal Spray
- Placebo Nasal Spray (Placebo Comparator): The placebo was administered via nasal inhalation with one spray in each nostril twice daily.
  Batch Number KL0781, Expiry Date Mar 2015.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Azelastine HCl and Fluticasone Propionate Nasal Spray, 137 µg/50 µg per spray — During the placebo lead-in period, the placebo nasal spray was administered via nasal inhalation with one spray in each nostril twice daily for 7days.
  During the randomized treatment period, the investigational products (experimental, active comparator and placebo nasal spray) were administered via nasal inhalation with one spray in each nostril twice daily for 14 days
  Arms: Azelastine HCl and Fluticasone Propionate Nasal Spray
Drug: Dymista™ Nasal Spray
  Arms: Dymista™ Nasal Spray
Drug: Placebo
  Arms: Placebo Nasal Spray

SUMMARY:
This study is to evaluate the equivalence of generic Azelastine Hydrochloride and Fluticasone Propionate Nasal Spray with that of the marketed drug, Dymista™ Nasal Spray, in the treatment of seasonal allergic rhinitis, and to evaluate the safety and tolerability of generic Azelastine Hydrochloride and Fluticasone Propionate nasal spray compared with Dymista™ nasal spray.

ELIGIBILITY:
Inclusion Criteria:

Subjects who met all of the following criteria were eligible for inclusion in the study:

1. Subjects who provided written informed consent.
2. Subjects who were able to read and understand English.
3. Males or females, 18 to 65 years old, inclusive.
4. If the subject was a female of childbearing potential, she was not pregnant (confirmed by negative urine pregnancy test) or lactating. Females of childbearing potential agreed to use reliable birth control measures throughout the study, defined as abstinence or use of an effective method of birth control (double barrier [female subject's partner using condom and female subject using diaphragm, contraceptive sponge, spermicide, or intrauterine device], or the use of a hormonal contraceptive [oral, patch, or inserted under the skin or injected into the muscle]). Female subjects who used oral contraceptives or levonorgestrel implants were required to have started the method at least 90 days prior to the screening visit. A female of childbearing potential was defined as a female who had experienced menarche, and who had not undergone successful surgical sterilization (hysterectomy, bilateral oophorectomy or ovariectomy, bilateral tubal ligation or salpingectomy) or was not post-menopausal for at least 1 year.
5. At least a 2-year reliable medical history consistent with SAR, defined as symptoms present during the previous two grass and/or pollen seasons.
6. Positive skin test within 12 months of screening to at least one currently present seasonal allergen in the geographical area that had a predictable allergen season (eg, birch pollen, ragweed, Mountain Cedar, etc) with a minimum skin test response of 3 mm or greater than a negative control, and a positive test to histamine, also defined as a response of 3 mm or greater than the negative control.
7. Was capable of tolerating intranasal application of the study drug.
8. No clinically significant results from the screening physical examination, nasal examination, and medical history.
9. Was willing and able to comply with the requirements of the protocol and was available for the full duration of the study, with no planned travel outside of the pollen area for a substantial portion (>48 hours) of the study period.
10. Was, in the Investigator's judgment (through exposure to allergen), expected to require treatment throughout the entire study period.

Exclusion Criteria:

Subjects who met any of the following criteria were excluded from the study:

1. Signs or symptoms of nasal polyps, deviated septum, or any other condition (including nasal piercing within the previous 3 months) which, in the opinion of the Investigator, may have resulted in erroneous study data.
2. Underwent nasal surgery or had nasal trauma within 3 months of Visit 1 (screening).
3. Had active respiratory conditions that included, but were not limited to, acute or exacerbated chronic sinusitis, an abnormal sinus radiograph, an upper or lower respiratory tract infection, or rhinitis medicamentosa.
4. Had PAR that required or was expected to require active PAR treatment during the study period.
5. Had a respiratory tract infection (including otitis media and streptococcus) that required antibiotic treatment within 2 weeks of Visit 1 (screening).
6. Used any of the prohibited medications prior to the start of the single-blind, placebo lead-in visit (Visit 2) within the time period specified in the protocol

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 595 (Actual)
Dates: Start 2013-12; Primary Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Treatment of Seasonal Allergic Rhinitis (Change from baseline in the combined reflective TNSS (combined AM and PM reflective scores of runny nose, nasal congestion, nasal itchiness, and sneezing) | 2 months
  Change from baseline in the combined AM and PM instantaneous scores of runny nose, nasal congestion, nasal itchiness, and sneezing.

SECONDARY OUTCOMES:
Treatment of Seasonal Allergic Rhinitis (Change from baseline in the combined AM and PM instantaneous scores of runny nose, nasal congestion, nasal itchiness, and sneezing.) | 2 months
  Change from baseline in the combined AM and PM instantaneous scores of runny nose, nasal congestion, nasal itchiness, and sneezing.